CLINICAL TRIAL: NCT01074346
Title: A Prospective, Multi-center, Observational Study to Assess the Tolerability of Interferon-beta 1-A (Rebif®) Therapy for Korean Patients With Multiple Sclerosis
Brief Title: Tolerability of Rebif® (Interferon-beta 1-A) Therapy in Korean Patients With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR 701068-511
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Interferon-beta 1-a
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Interferon-β-1a — Interferon-β-1a according to the standard practice
  Other Names: Rebif®

SUMMARY:
This is an observational study to assess the tolerability of Rebif treatment in Korean multiple sclerosis (MS) subjects.

DETAILED DESCRIPTION:
The present observational study is being conducted to assess the safety information from a target of 100 Korean subjects with MS treated with Rebif. Various parameters like subjects' background (age, sex, BMI), MS history, MS status (MS type, Expanded Disability Status Score [EDSS] and others), MS Treatment Concern Questionnaire (MSTCQ), Rebif treatment status, concomitant disease modifying agents (DMA) therapy and Rebif related adverse events will be collected. Subjects will be followed for 12 months. Proportion of subjects with moderate to severe (Grade 3-5) injection site reactions after 3, 6, 12 months of Rebif treatment will be determined. Secondary outcomes like annual relapse rate, change in EDSS, changes in MSTCQ, time to first relapse and incidence of side effects associated with Rebif therapy will also be determined and presented descriptively.

OBJECTIVES

Primary objectives

* To assess the tolerability of Rebif treatment in Korean MS subjects in a non-interventional setting Secondary Objectives
* To evaluate subject's satisfaction, clinical data and disease characteristics of the population of MS subjects undergoing Rebif treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, who are eligible for Rebif treatment according to the indication in the national label of Rebif in Korean subjects with MS. The national labels approved by Korean Regulatory Authority are:

  1. Subjects with relapsing MS with two or more acute exacerbations in the previous two years
  2. Subjects with secondary progressive MS with ongoing relapsing activity
* Subjects who sign the informed consent form.

Exclusion Criteria:

* Initiation of treatment in pregnancy.
* Subjects with a history of hypersensitivity to natural or recombinant interferon-ß, or to any excipients.
* Subjects with current severe depression and/or suicidal ideation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with MS undergoing treatment with Rebif in Korea.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with moderate to severe (grade 3-5) injection site reactions based on pain, bruising and/or transient (<24 hours) erythema; inflammation alone and with induration; necrosis at injection site; plastic surgery required for necrosis | After 3, 6 and 12 months of Rebif treatment

SECONDARY OUTCOMES:
Annual relapse rate | Baseline to 12 months observation period
Change in EDSS | Baseline to 12 months observation period
Change in MSTCQ | Baseline to 12 months observation period
Time to first relapse | Baseline to 12 months observation period
Incidence of side effects associated with Rebif therapy | Baseline to 12 months observation period

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, 50 Ilwon-dong, Gangnam-gu, South Korea